CLINICAL TRIAL: NCT04211220
Title: Clinical Evaluation of Insulin Real-Time Advisor (IRTA©): a Decision Support Software for Insulin Therapy Combined With Freestyle Libre®, a Continuous Glucose Monitoring System: Glycemic Impact and Satisfaction in Type 1 Diabetic Patients
Brief Title: Study to Assess the Metabolic Impact of IRTA© and Patients Satisfaction in Type 1 Diabetic Patients, Treated by Either Insulin Pump or Multiple Daily Insulin Injections, and Using Freestyle Libre®, a Real-time Continuous Glucose Monitoring
Acronym: IRTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC19_8858_IRTA
Record Dates: First submitted 2019-12-20; First posted 2019-12-26 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
Keywords: Real time continuous glucose monitoring; Decision support software
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A decision support software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 1 diabetes (Experimental)
  Interventions: Other: A decision support software

INTERVENTIONS:
Other: A decision support software — Insulin pump Continuous glucose monitoring

SUMMARY:
A prospective monocentric " before and after " study, ruled in 2 periods of 3 months : during the first period, the patient will adjust insulin treatment as usual, during the second period, the patient will adjust insulin treatment with IRTA support

DETAILED DESCRIPTION:
Freestyle Libre® continuous glucose monitoring (CGM) system may improve glycemic control. However, this system contributes to the complexity of insulin adjustment by the diversity of the data delivered by CGM system.

Insulin Real-Time Advisor (IRTA©), a decision support software, has been developed in order to guide patients in the adaptation of their treatment according to CGM data. IRTA© provides advice applicable to thousand situations according to six parameters: glucose level, trend arrows, meals, physical activity, before bedtime, time since the previous bolus.

Type of advice :

* Insulin injection (carb and correction)
* To continue treatment without modification
* To lower the insulin dose (temporary basal rate)
* Sugar intake advice
* Glucose level control with CGM, self-monitor blood glucose, blood ketones monitor
* To change catheter for patients treated by insulin pump.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Patients with type 1 diabetes mellitus for more than 2 years
* Treated by either insulin pump for more than 6 months or multiple daily insulin injections.
* Using Freestyle Libre® for more than 3 months
* Accepting IRTA use
* Patient able to provide free and informed consent
* Patient able to provide written non-disclosure agreement

Exclusion Criteria:

* Pregnancy, breastfeeding or pregnancy project in the future 6 months
* Patients with no smart phone or internet access
* Patients legally protected (under judicial protection, guardianship or supervision)
* Patients with acute illness (psychiatric, infection, cancer,…)
* Patients using another CGM system (Enlite® or Dexcom G4®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in 70-180mg/dl (time in range) in the last month of each period of the study (without and then with IRTA©) | 6 months
  Assessment of the metabolic impact of IRTA© on "time in range" (time spent in the standard glucose range between 70-180mg/dl, ie 3.9-10mmol/l) in type 1 diabetic patients, treated by either insulin pump or multiple daily insulin injections, and using Freestyle Libre®.

SECONDARY OUTCOMES:
Comparison of HbA1c level at the end of each period of the study (without / with IRTA©) | 6 months
  Blood sample at inclusion, 3 months and 6 months
Time spent in glucose level higher than 250 mg/dl | 6 months
Time spent in glucose level higher than 180 mg/dl | 6 months
Time spent in glucose level lower than 70 mg/dl | 6 months
Time spent in glucose level lower than 54 mg/dl | 6 months
Number of incidents (severe hypoglycemia, diabetic ketoacidosis, hospitalizations related to poor glycemic control) | 6 months
Percentage of time spent with or without CGM | 6 months
Glycemic variability | 6 months
Patients' satisfaction related to CGM and the impact of IRTA© on this satisfaction | 6 months
  CGM Satisfaction (CGM-SAT) 44-item questionnaire. Higher scores reflect more favorable impact of, and satisfaction with, CGM use.
Patients' satisfaction related to IRTA© | 6 months
  Satisfaction questionnaire: 5-point Likert scale (1 = strongly agree; 5 = strongly disagree) with each of 18 items.
Number of connections to the IRTA system | 6 months
Number of advice given by the IRTA system | 6 months
Type of advice given by the IRTA system that is more often asked | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No